CLINICAL TRIAL: NCT00005411
Title: Study of Children's Activity and Nutrition (SCAN)--Extended Analyses
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4329; R03HL047388 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-03

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Coronary Heart Disease Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases

SUMMARY:
To continue analysis of data from a longitudinal study of 246 urban Black preschool children and their families in order to identify the long-term effects of social and environmental influences on nutrition and activity and the consequences of these influences for the children's cardiovascular disease (CVD) risk status.

DETAILED DESCRIPTION:
BACKGROUND:

This study contributed to understanding the development of patterns of eating and exercise, focusing on environmental influences that promoted healthful life styles and prevented risk behaviors for CVD.

DESIGN NARRATIVE:

The data set included additional measures of activity and nutrition of the preschool child as well as measures of the activity of an older sibling and mother. The data were gathered in the homes and schools of the children and included both self-report and direct measurement of activity and nutrition. Additional assessments of activity, lipid fractions and apolipoproteins, and Type A Behavior Patterns and Life Stress in the preschool child, i.e., target child , an older sibling and the children's mother added considerably to the complexity and value of the data set permitting additional questions regarding the development of activity, the influences of siblings and parents on this development, and the relationship to CVD risk status and Type A Behavior Patterns.

Hypotheses addressed included 1. Activity levels and the activities selected showed increasing stability with age in preschool and older Black children. 2. The influence of parental prompts and family environment on activity increased asymptotically with age: The effects increased during early childhood; the effects did not increase significantly in older children. 3. Older sibling's influence on the target child's behavior increased with age. The target child's CVD risk status became more like the older sibling's with age. 4. Perceptions of recent Life Stress and ratings of Type A Behavior Patterns for target child, the older sibling, and mother were predisposing variables that were positively related to the target child's activity. 5. Long-term patterns of physical activity were associated with HDL and apo A-1 in the target child and the older sibling; the effect was stronger for the older sibling. Long-term patterns of the target child's nutrient intake were associated with his/her lipid levels.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-09; Study Completion 1993-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Iannotti — Georgetown University

REFERENCES:
- [Background] Iannotti RJ, Zuckerman AE, Blyer EM, O'Brien RW, Finn J, Spillman DM. Comparison of dietary intake methods with young children. Psychol Rep. 1994 Jun;74(3 Pt 1):883-9. doi: 10.2466/pr0.1994.74.3.883. PMID 8058872
- [Background] Iannotti RJ, O'Brien RW, Spillman DM. Parental and peer influences on food consumption of preschool African-American children. Percept Mot Skills. 1994 Oct;79(2):747-52. doi: 10.2466/pms.1994.79.2.747. PMID 7870497